CLINICAL TRIAL: NCT00649896
Title: Comparative Evaluation of the Adhesion Quality of a New Formulation of the Mylan Estradiol Transdermal System (0.025 mg/Day; Mylan) and Climara® Transdermal System (0.025 mg/Day; Berlex) in Healthy Postmenopausal Female Volunteers
Brief Title: Evaluation of Adhesion Quality of a New Formulation of the Mylan Estradiol Transdermal System 0.025 mg/Day and Climara® Transdermal System 0.025 mg/Day
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mylan Pharmaceuticals Inc (Industry)
Responsible Party: Will Sullivan, Global Head of Product Risk and Safety Management, Mylan Inc.
Organization: MylanPharma (Unknown)
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: ESTR-0334
Record Dates: First submitted 2008-03-30; First posted 2008-04-01 (Estimated); Last update posted 2008-04-01 (Estimated); Status verified 2008-03

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- 1 (Experimental): Mylan Estradiol Transdermal System 0.025 mg/day
  Interventions: Drug: Mylan Estradiol Transdermal System 0.025 mg/day
- 2 (Active Comparator): Climara® Transdermal System 0.025 mg/day
  Interventions: Drug: Climara® Transdermal System 0.025 mg/day

INTERVENTIONS:
Drug: Mylan Estradiol Transdermal System 0.025 mg/day
  Arms: 1
Drug: Climara® Transdermal System 0.025 mg/day
  Arms: 2

SUMMARY:
The primary objective of this study was to compare the adhesive quality of a new formulation of the Mylan Estradiol Transdermal System with that of Climara® Transdermal System following a single system application in 80 healthy postmenopausal female volunteers. As a secondary objective, primary dermal irritation was assessed after removal of each transdermal system.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 40-69 years.
2. Sex: Females only.
3. Weight: At least 52 kg (115 lbs) and within 30% of Ideal Body Weight (IBW), as referenced by the Table of "Desirable Weights of Adults" from Metropolitan Life Insurance Company, 1999 (See Part II: ADMINISTRATIVE ASPECTS OF HUMAN BIOAVAILABILITY PROTOCOLS).
4. Absence of menses for one year for postmenopausal subjects, or at least 6 weeks for oophorectomized subjects. (For oophorectomized subjects, an operative report documenting bilateral oophorectomy and surgical pathology report documenting the absence of malignant disease.)
5. Baseline FSH and 17-beta-estradiol serum levels consistent with postmenopausal status confirmed within 14 days of initiation of study medication. (FSH greater than or equal to 40 mIU/mL; 17-beta-estradiol less than or equal to 31 pg/mL)
6. All subjects should be judged normal and healthy during a prestudy medical evaluation (physical examination, laboratory evaluation and 12-lead ECG) performed within 14 days of the initial patch application.
7. The physical examination shall include pelvic and breast exams.

   a. Pelvic findings should be consistent with hypoestrogenemia. b. A mammogram will be required if not performed within the last 12 months. c. A Papanicolaou ("Pap") smear will be required on subjects with an intact uterus and cervix if not performed within the last 6 months.

Exclusion Criteria:

1. Institutionalized subjects will not be used.
2. Social Habits:

   a. Use of any tobacco products. b. Ingestion of any alcoholic, caffeine- or xanthine-containing food or beverage within the 48 hours prior to the initial dose of study medication.

   c. Ingestion of any vitamins within the 48 hours prior to the initial dose of study medication.

   d. Any recent, significant change in dietary or exercise habits.
3. Medications:

   1. Use of any medication within 14 days prior to the initial dose of study medication.
   2. Use of any medication known to alter hepatic enzyme activity within 28 days prior to the initial dose of study medication.
   3. Use of any systemic antibiotics, estrogens, or hormones within 28 days prior to the initial dose of study medication.
4. Diseases:

   1. History of any significant chronic disease such as (but not limited to):

1. Thrombotic disorders. 2. Coronary artery or cerebrovascular disease. 3. Liver, kidney or gallbladder dysfunction/disorder(s). 4. Fibrocystic disease or breast nodules. 5. Family history of breast cancer. 6. Diabetes or any other endocrinological disease. 7. Estrogen-dependent neoplasia. 8. Postmenopausal uterine bleeding. 9. Endometrial hyperplasia. b. History of drug and/or alcohol abuse. c. Acute illness at the time of either the prestudy medical evaluation or dosing.

5. Abnormal and clinically significant laboratory test results:

1. Clinically significant deviation from the Guide to Clinically Relevant Abnormalities (See Part II: ADMINISTRATIVE ASPECTS OF BIOEQUIVALENCE PROTOCOLS).
2. Abnormal and clinically relevant ECG tracing. 6. Subjects who have received an investigational drug within 30 days prior to the initial dose of study medication.

   7. Allergy or hypersensitivity to tapes or adhesives (ex. Band-aids, medical tape), estradiol or other hormonal products.

Ages: 40 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2003-08; Primary Completion 2003-09 (Actual); Study Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
Dermal Safety | within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence A Galitz, M.D., Principal Investigator — SFBC International
Locations (1):
- SFBC International, Miami, Florida, United States

REFERENCES:
- See also: Mylan Pharmaceuticals Inc. - Clinical Trial Results — http://www.mpibiostudies.com
- See also: Daily Med - posting of most recent submitted labelling to the Food and Drug Administration (FDA) and currently in use — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.html